CLINICAL TRIAL: NCT03001167
Title: Early Life Antibiotics, Gut Microbiome Development, and Risk of Childhood Obesity
Brief Title: Microbiome, Antibiotics, and Growth Infant Cohort
Acronym: MAGIC
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Minnesota (Other); University of Pennsylvania (Other); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 15-012623; R01AI121383 (NIH)
Record Dates: First submitted 2016-12-15; First posted 2016-12-22 (Estimated); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Obesity, Childhood; Antibiotic Side Effect
Keywords: Microbiome; Antibiotics; Growth
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples Saliva samples nasal swab skin swabs blood draw cord blood heel stick
Oversight: Data Monitoring Committee: No

SUMMARY:
This cross-disciplinary study will assemble and longitudinally follow a large, diverse birth cohort to determine the relationships between early life antibiotic exposure, microbiome development, growth, antibodies, and immunostimulation.

DETAILED DESCRIPTION:
Perinatal and infant antibiotic exposures are common and have been linked to changes in the gut microbiome, which plays a central role in health and disease. Childhood obesity is an epidemic and animal models have linked antibiotic induced changes in the microbiome with increased adiposity. Infants become colonized with trillions of bacteria in the first few hours of life. During this time period, their nascent immune system develops tolerance to commensal microbes

The primary objectives are to measure the impact of common perinatal and early childhood antibiotic exposures on the structure and function of the developing gut microbiome. To determine the association between common perinatal and early childhood antibiotic exposures and weight/adiposity gain in a large birth cohort of children. To determine mechanisms for the association between microbiome changes over time and the rate of weight/adiposity gain in a large birth cohort of children. To determine the normal developmental pattern by which healthy children develop antibodies in their blood against the microbes that naturally colonize their intestines. To determine the association between immunostimulation and protection from persistent colonization in humans.

ELIGIBILITY:
Inclusion Criteria (if not specified, applies to child):

* Born at Pennsylvania Hospital
* Recruited at <120 hours of age
* Born at ≥36 0/7 weeks gestation
* Birth weight ≥2000 grams
* Parents plan to receive well-child care in the Children's Hospital of Philadelphia (CHOP) network, Society Hill Pediatrics, Center City Pediatrics, Penn Medicine or South Philly Pediatrics
* Biological mother is the legal guardian, or the child is born from a surrogacy with guardianship immediately transferred in hospital

Exclusion Criteria (if not specified, applies to child):

* Child in neonatal intensive care unit (NICU) for >120 cumulative hours
* Biological mother NOT legal guardian, except surrogacy where guardianship is transferred at birth
* Biological mother NOT primary caretaker, except surrogacy where guardianship is transferred at birth
* Biological mother < 18 years of age
* Child has culture confirmed (blood or cerebrospinal fluid cultures) infection
* Biological mother is non-English speaking

Max Age: 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Our study population will be comprised of children born at Pennsylvania Hospital between 2016-2018 and subsequently, followed in the Children's Hospital of Philadelphia (CHOP) Care Network or one of four other local primary care pediatric practices.
Sampling Method: Non-Probability Sample
Enrollment: 509 (Actual)
Dates: Start 2016-12-09 (Actual); Primary Completion 2021-10-22 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
cumulative microbial diversity | 24 months
weight trajectory adjusted for time varying length | 24 months

SECONDARY OUTCOMES:
total number of individual bacterial taxa | 24 months
expression levels of bacterial gene categories | 24 months
fat stores in the upper arm/extremity | 24 months
  Skinfolds at the triceps are measured (0.1 mm) with a skinfold caliper
fat stores in the upper back/trunk | 24 months
  Skinfolds at the superiliac and subscapular sites are measured (0.1 mm) with a skinfold caliper
supine length trajectory | 24 months
determine the association between immunostimulation and protection from persistent colonization in humans | 24 months
Use autologous serum antibodies to "tag" fecal microbes | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey S Gerber, MD, PhD, Principal Investigator — Children's Hospital of Philadelphia; Dan Knights, PhD, Principal Investigator — University of Minnesota
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data will be shared with collaborators at the Knights Lab at the University of Minnesota.

REFERENCES:
- See also: Official study website — https://magicstudy.research.chop.edu/